CLINICAL TRIAL: NCT04264364
Title: Endoscopic Sleeve Gastroplasty in Comparison With Laparoscopic Sleeve Gastrectomy in Terms of Short-Term Nutritional Outcomes
Brief Title: ESG vs LSG: Short-term Nutritional Outcomes
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Collaborators: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Ghadah AlGhafees, Clinical Nutrition Master's Student, King Saud University
Other Study IDs: ESGvsLSG
Record Dates: First submitted 2020-01-30; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Endoscopic Sleeve Gastroplasty; Laparoscopic Sleeve Gastrectomy; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic sleeve gastrectomy: Patients who underwent laparoscopic sleeve gastrectomy
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- endoscopic sleeve gastroplasty: Patients who underwent endoscopic sleeve gastroplasty
  Interventions: Procedure: Endoscopic sleeve gastroplasty

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Bariatric surgical intervention
  Groups: laparoscopic sleeve gastrectomy
Procedure: Endoscopic sleeve gastroplasty — Endoscopic bariatric procedure
  Groups: endoscopic sleeve gastroplasty

SUMMARY:
To assess endoscopic sleeve gastroplasty in comparison to laparoscopic sleeve gastrectomy before and 3 months after the procedure in terms of multiple nutrition-related factors, quality of life, weight and other related parameters.

DETAILED DESCRIPTION:
This will be a short-term prospective cohort study, single-center study (NewYou clinical center - Riyadh). A total of 15 endoscopic sleeve gastroplasty patients will be matched with 15 laparoscopic sleeve gastrectomy patients by age, gender and BMI. Total sample size is 30 patients. Sample size was selected based on literature, considering the sample will be surgical patients and based on booked patients in the clinic. A multidisciplinary team will provide post-procedure care (including post-surgery diet stages protocol given by the center).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old)
* Willingness and ability to participate
* Males and females
* Non-pregnant

Exclusion Criteria:

* Children (<18 years old)
* Pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 27 LSG patients 30 ESG patients
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 3 months
  Weight Loss in kilograms (baseline weight in kilogram - follow-up weight in kilogram)
Percentage of total weight loss (%TWL) | 3 months
  %TWL = [(baseline weight in kilogram - weight at 3 months in kilogram) ÷ baseline weight in kilogram]
Percentage of excess weight loss (%EWL) | 3 months
  %EWL = [percentage of weight lost compared with excess weight, which is defined as baseline weight in kilogram - the weight corresponding to a BMI of 25 kg/m^2 in kilogram])
Waist Circumference | 3 months
  Waist Circumference in centimeters
body fat percentage change | 3 months
  change in body fat percentage between baseline and follow-up visits as calculated by a calibrated bioelectrical impedance device
fat mass change | 3 months
  change in fat mass in kilograms between baseline and follow-up visits as calculated by a calibrated bioelectrical impedance device
fat mass index change | 3 months
  change in fat mass index in kg/m^2 between baseline and follow-up visits as calculated by a calibrated bioelectrical impedance device
fat free mass change | 3 months
  change in fat free mass in kilograms between baseline and follow-up visits as calculated by a calibrated bioelectrical impedance device
fat free mass index change | 3 months
  change in fat free mass index in kg/m^2 between baseline and follow-up visits as calculated by a calibrated bioelectrical impedance device
skeletal muscle mass change | 3 months
  change in skeletal muscle mass in kilograms between baseline and follow-up visits as calculated by a calibrated bioelectrical impedance device
Dietary habits | 3 months
  Assessment of dietary habits using the How Healthy Is Your Diet questionnaire, developed by the British Heart Foundation 2012
  The score is from 0 minimum to 29. Higher score correlates with better dietary habits.
24-hour dietary recall | 3 months
  Assessment of nutritional intake with 24-hour dietary recall form
3-day dietary record | 3 months
  Assessment of nutritional intake with 3-day dietary record
Change in quality of life after procedure | 3 months
  Moorehead-Ardelt Quality of Life Questionnaire II scoring using Moorehead-Ardelt Quality of Life Questionnaire II Self Esteem and Activity Levels SCORING KEY minimum score is -3 and maximum score is 3 a higher score means a better outcome.
Cholesterol Biochemical assessment (laboratory assessment) | 3 months
  Cholesterol in milligrams per deciliter (< 200 Desirable)
Alanine Aminotransferase Biochemical assessment (laboratory assessment) | 3 months
  Alanine Aminotransferase in units per liter (up to 33)
Gamma glutamyl transferase Biochemical assessment (laboratory assessment) | 3 months
  Gamma glutamyl transferase in units per liter (< 40)
sodium Biochemical assessment (laboratory assessment) | 3 months
  sodium in millimoles/liter (136-145)
platelets Biochemical assessment (laboratory assessment) | 3 months
  platelets in cmm (150.0-450.0)
MCH Biochemical assessment (laboratory assessment) | 3 months
  MCH in picograms per cell (25.00-32.00)
potassium Biochemical assessment (laboratory assessment) | 3 months
  potassium in millimoles/liter (3.5-5.1)
MCV Biochemical assessment (laboratory assessment) | 3 months
  MCV in femtoliters per cell (76.00-97.00)
MCHC Biochemical assessment (laboratory assessment) | 3 months
  MCHC in grams per deciliter (31.80-35.40)
Chloride Biochemical assessment (laboratory assessment) | 3 months
  Chloride in millimoles/liter (97-111)
creatinine Biochemical assessment (laboratory assessment) | 3 months
  creatinine in mg/dL (44-80)
WBC Biochemical assessment (laboratory assessment) | 3 months
  WBC in × 10^9/L (4.00-11.00)
RBC Biochemical assessment (laboratory assessment) | 3 months
  RBC in million mcL (3.80-5.80)
HCT Biochemical assessment (laboratory assessment) | 3 months
  HCT in % (36.00-46.00)
serum glucose Biochemical assessment (laboratory assessment) | 3 months
  serum glucose in mg/dL (70-150)
serum TSH Biochemical assessment (laboratory assessment) | 3 months
  serum TSH in milli-international units per liter (0.38-5.33)
hemoglobin Biochemical assessment (laboratory assessment) | 3 months
  hemoglobin in grams per deciliter (12.00-16.00)
Eosinophils Biochemical assessment (laboratory assessment) | 3 months
  Eosinophils in cells per microliter (0.00-6.00)
monocytes Biochemical assessment (laboratory assessment) | 3 months
  monocytes in percent (0.00-13.70)
INR plasma ratio Biochemical assessment (laboratory assessment) | 3 months
  INR plasma ratio (no units)
Basophils Biochemical assessment (laboratory assessment) | 3 months
  Basophils in basophils per microliter (0.00-1.00)
MPV Biochemical assessment (laboratory assessment) | 3 months
  MPV in fl (7.20-11.10)
RDW Biochemical assessment (laboratory assessment) | 3 months
  RDW in % (12.40-16.20)
lymphocytes Biochemical assessment (laboratory assessment) | 3 months
  lymphocytes in % (15.00-50.00)
neutrophils Biochemical assessment (laboratory assessment) | 3 months
  neutrophils in cells/µL (40.00-75.00)

CONTACTS AND LOCATIONS:
Overall Officials: Ghadah M AlGhafees, BSc, Principal Investigator — King Saud University
Locations (1):
- New You Medical Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided